CLINICAL TRIAL: NCT07304115
Title: Noise Associated With a Mechanical Heart Valve Prosthesis: Does the Memory of Preoperative Information Have an Influence on Postoperative Quality of Life?
Acronym: QUALICLIC
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240701; 2024-A01122-45 (Other: ANSM)
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Mechanical Heart Valve Prosthesis
Keywords: mechanical heart valve prosthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an aortic mechanical valve who have consulted at the Marfan reference center: All adult patients with an aortic mechanical valve who have consulted at the Marfan reference center

SUMMARY:
As part of the follow-up in the Day Hospital in the national reference center for Marfan syndrome and related disorders, each consultant benefits from a psychological interview.

During these psychological interviews, it is noticed that some patients with a mechanical heart valve prosthesis are bothered on a daily basis by the noise caused by this valve. Some patients also mention the fact that the noise of their mechanical heart valve prosthesis causes discomfort to their partners.

Indeed, preoperatively to aortic surgery, the need for aortic valve replacement is evaluated and the patient must receive a clear and detailed explanation of the advantages and disadvantages associated with a mechanical heart valve prosthesis and a biological heart valve prosthesis so that he or she can make an informed choice.

Nevertheless, during their psychological interviews, it was noted that the memory of the information concerning the noise associated with mechanical heart valve prostheses is not systematically delivered preoperatively. While there are studies in the literature showing that the noise of the mechanical valve prosthesis has harmful consequences on the quality of life and sleep of the patient and/or those around them, no study has determined whether giving information on the noise associated with the mechanical valve preoperatively will have consequences on the post-operative quality of life of the patient and those around them.

DETAILED DESCRIPTION:
During cardiac surgery in people with Marfan Syndrome, it is not uncommon for an aortic or mitral valve replacement to be performed. Several types of valve substitutes exist, each with its advantages and disadvantages: biological valve prostheses made with animal tissue and mechanical valve prostheses made of synthetic materials (pyrolytic carbon and titanium) are mainly implanted.

Heart valve surgery is necessary on average before the age of 40 in Marfan syndrome, i.e. at a younger age than in other heart valve pathologies.

The recommendations are to prefer a mechanical valve prosthesis in subjects under 60 years of age because these mechanical prostheses have a longer lifespan than biological prostheses, especially in young subjects. However, the implantation of a mechanical valve prosthesis has two main disadvantages compared to the biological prosthesis:

1. the need to take anticoagulant treatment with Anti Vitamin K for life
2. the noise generated by the wings of the mechanical prosthesis when they close

Data from the literature confirm that this noise is potentially harmful to patients' quality of life, since one to three-quarters of patients are regularly bothered by the noise generated by the mechanical prosthesis and that this noise can disturb patients during the day but also during their sleep. However, it appears that most patients are not informed preoperatively that a mechanical prosthesis generates a noise that they will be able to hear.

A study that involved nearly 1200 patients with mechanical prostheses reported that valve noise is felt more negatively in women and patients under 60 years of age.

Based on data from the literature, it appears that the noise generated by mechanical valves can be harmful to some patients and impact the quality of life of some patients.

On the other hand, the frequency and effect on quality of life of providing information to the patient preoperatively on the advantages and disadvantages of the different types of valve replacement has not been studied, or very little.

This study wants to determine whether the recall of preoperative information about the noise caused by the mechanical valve has consequences on the postoperative quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an aortic mechanical valve who have consulted from 1995 to date at the reference center.
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Patient who does not speak French
* Hearing or hearing impaired patient.
* Patient without a phone: Interviews will take place over the phone.
* Patient who has been individually informed and objects to participate in this research
* Patient not affiliated to a social security scheme or CMU (Universal health coverage)
* Adult patients protected by law
* Patient on AME (State medical aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of legal age and implanted with an aortic mechanical valve.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative quality of life assessed by the answers to the SF36 questionnaire | 1 year
  To determine whether the recall of preoperative information about the noise caused by the mechanical valve has consequences for patients' postoperative quality of life.

SECONDARY OUTCOMES:
Gender (male) | 1 year
  Determine whether being a male is a determinant of discomfort related to mechanical valve noise.
Gender (female) | 1 year
  Determine whether being a female is a determinant of discomfort related to mechanical valve noise.
Percentage of patients who would have chosen not to receive mechanical valves | 1 year
  To determine whether recalling preoperative noise information would have changed the patient's choice of valve replacement type.
Operation in an emergency | 1 year
  Comparison between patients who were operated on in an emergency and those who were operated on during scheduled surgery to determine the impact of emergency surgery compared to scheduled surgery on the discomfort caused by mechanical valve noise.
Scheduled surgery | 1 year
  Comparison between patients who were operated on in an emergency and those who were operated on during scheduled surgery to determine the impact of emergency surgery compared to scheduled surgery on the discomfort caused by mechanical valve noise.
Patients who were operated on before 2004 | 1 year
  Comparison to determine whether there is a significant difference in responses between patients who have had surgery more than 20 years ago (before the year 2004) and those who have had surgery in the last 20 years.
Patients who were operated on after 2004 | 1 year
  Comparison to determine whether there is a significant difference in responses between patients who have had surgery more than 20 years ago (before the year 2004) and those who have had surgery in the last 20 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: No